CLINICAL TRIAL: NCT04463030
Title: Clinical Pilot Study on Antioxidant Uptake and Downstream Effects
Brief Title: Antioxidant Bioavailability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Principal Investigator, Gitte Jensen, Ph.D., Research Director, Natural Immune Systems Inc
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NIS161-004
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, single blind, cross-over trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Liposomal vitamin C, 1 gram (Active Comparator): Participants will consume 1 gram on study day
  Interventions: Dietary Supplement: Liposomal vitamin C, 1 gram
- Liposomal vitamin C, 2 grams (Active Comparator): Participants will consume 2 grams on study day
  Interventions: Dietary Supplement: Liposomal vitamin C, 2 grams
- Liposomal vitamin C, 5 grams (Active Comparator): Participants will consume 5 grams on study day
  Interventions: Dietary Supplement: Liposomal vitamin C, 5 grams
- Placebo (Placebo Comparator): Participants will consume placebo on study day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Liposomal vitamin C, 1 gram — after a blood draw 1 gram of vitamin c will be consumed followed by 3 additional blood draws
  Arms: Liposomal vitamin C, 1 gram
Dietary Supplement: Liposomal vitamin C, 2 grams — after a blood draw 2 grams of vitamin c will be consumed followed by 3 additional blood draws
  Arms: Liposomal vitamin C, 2 grams
Dietary Supplement: Liposomal vitamin C, 5 grams — after a blood draw 5 grams of vitamin c will be consumed followed by 3 additional blood draws
  Arms: Liposomal vitamin C, 5 grams
Dietary Supplement: Placebo — after a blood draw placebo will be consumed followed by 3 additional blood draws
  Arms: Placebo

SUMMARY:
A small cross-over trial on 3 different doses of liposomal vitamin C, comparing vitamin C uptake and downstream effects when 24 people consume 1, 2, and 5 grams on different test days, compared to placebo.

DETAILED DESCRIPTION:
A randomized, cross-over study design will be used to evaluate the effects of consumption of 4 different doses of liposomal vitamin C (0, 1, 2, and 5 grams). The study is of 5 weeks' duration, with evaluation of a different dose at each of week 1, week 3 and week 5 with a one week washout between each dose.

ELIGIBILITY:
Inclusion Criteria:

* Adult people of either gender;
* BMI between 18.0 and 34.9 (inclusive);
* Willing to abstain from coffee, tea, and soft-drinks for at least one hour prior to a clinic visit;
* Willing to abstain from alcohol for at least 12 hours prior to a clinic visit;
* Willing to maintain a consistent habit of abstaining from exercising, tobacco use, and nutritional supplements on the morning of a study visit.

Exclusion Criteria:

* Cancer during past 12 months;
* Chemotherapy during past 12 months;
* Significant active uncontrolled illness (such as lymphoma, liver disease, kidney failure, heart failure).
* Previous major surgery to stomach or intestines [(absorption of test product may be altered) minor surgery is not a problem, including appendix and gallbladder removal];
* Currently taking nutritional supplements judged by the study coordinator to negate or camouflage the effects of the test product;
* Food allergies related to ingredients in test product;
* Women who are pregnant, nursing, or trying to become pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-06-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of vitamin C levels | 6 hours
  HPLC (High performance liquid chromatography)

SECONDARY OUTCOMES:
Evaluation of antioxidant status | 6 hours
  FRAP (Ferric reducing antioxidant power) assay

OTHER OUTCOMES:
Evaluation of downstream effects reflecting antioxidant protection | 6 hours
  lipid peroxidation

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Jensen, PhD, Principal Investigator — NIS Labs
Locations (1):
- Gitte Jensen, Klamath Falls, Oregon, United States